CLINICAL TRIAL: NCT04352829
Title: THE EFFECT OF REPEATED VIDEO-TRAINING-SESSION ON METERED DOSE
Brief Title: VIDEO-TRAINING-SESSION ON METERED DOSE INHALER SKILLS AMONG INDIVIDUALS WITH COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, EBRU YILDIZ, lecturer, Mersin University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: VIDEO-TRAINING
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, metered dose inhaler, training nursing, video session
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: STUDY TYPE and STUDY AIM The study was experimentally undertaken in pre-test post-test control group design in order to assess the effect of video-training-session method upon adequacy of metered dose inhaler (MDI) among individuals with COPD.
  STUDY POPULATION and SAMPLING In case of drop outs (wish to withdraw from the study, early hospital discharge, loss of life, etc), 20 patients were assigned to each group. The first 20 COPD patients who met the inclusion criteria were assigned to the control group whereas the second 20 COPD patients were assigned to the experimental group.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPERİMENTAL GROUP (Experimental): 1st day, patients were asked to use an MDI sample that didn't contain an active agent. At the same time, they filled the MDI Skill Evaluation Form, obtaining 'the scores of the 1st measurement'. Next, MDI use was explained through the video twice. After each video and explanation, the patients were asked to use the same MDI sample for 10 min. Simultaneously, the skills were marked by the researcher through observation on the form, obtaining 'the scores of the 2nd measurement'. 2nd day, they were again asked to use the MDI. While using the MDI, the form was marked and 'the scores of the 3rd measurement' were found. Later, a video session was held as on the 1st day, the video was watched twice, and after each repetition, were requested to use the MDI again. While they were using the MDI, the skills were simultaneously marked on the form and 'the scores of the 4th measurement were determined. 3rd day, all steps were repeated.
  Interventions: Other: VIDEO-TRAINING-SESSION ABOUT MDI USE
- CONTROL GROUP (No Intervention): 20 patients were recruited to the control group. The controls received a routine training on MDI from their clinic nurses including verbal explanation of MDI use. The controls received training about MDI use in line with ethical principles and watched the video once after the 5th measurement. After the study, participants who wished to watch the training video again were provided internet links.

INTERVENTIONS:
Other: VIDEO-TRAINING-SESSION ABOUT MDI USE — The steps were demonstrated with the brochure that illustrated correct inhalation techniques and were prepared by Turkish Respiratory Research Society-Inhalation Treatment Study Group in line with the literature and were described with a video that was designed by Turkish National Society of Allergy and Clinical Immunology (25). The video is provided with a free access on the webpage of Turkish National Society of Allergy and Clinical Immunology.The video included images that explained the steps about what to do before MDI use, how to use the device and the issues to which attention should be paid during the use of the device and focused on the skill-steps that should gradually be performed about MDI use.
  Arms: EXPERİMENTAL GROUP

SUMMARY:
OBJECTIVE: This study was undertaken to assess the effect of repeated video-training sessions on the adequacy of metered-dose inhaler (MDI) among individuals with COPD.

BACKGROUND: MDI devices facilitate the use of inhalation drugs in COPD patients and have become ever more important over the years. However, this device requires a certain level of hand-to- mouth coordination and cognitive ability. Since it has a high risk of application errors, training in its use is important to treatment success.

DESIGN: Randomised controlled trial METHOD: This study was carried out from 1 February to 1 July 2017 with the participation of 40 COPD patients. The data were collected using a 'Patient Information Request Form' and an 'MDI Skill Evaluation Form'. CONSORT checklist was used to report the current study. RESULTS: It was found that there was no significant difference between the experimental and control groups in terms of the mean scores of the 1st measurement (p > .05), though the mean scores of the 5th measurement were significantly higher in the experimental group (p< .001). In the 5th measurement, it was identified that the control group had 'moderate' adequacy (3.20±1.6), while the experimental group had 'satisfactory' adequacy (8.70 ± 1.17), indicating that the patients in the experimental group made fewer mistakes and showed improved adequacy.

CONCLUSION: It was found that repeated video-training sessions materially improved MDI skills. Relevance to clinical practice. Supporting the training on inhaler drug therapy with visual technological tools and regular checking of drug use will contribute to COPD management.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) -one of the most important chronic health problems of respiratory system- is irreversible, progresses slowly and is characterized with chronic inflammation and airflow obstruction (1,2,3,4). According to the report of World Health Organization (WHO) "Non-communicable Diseases Progress Monitor 2017"; mortality rate in Turkiye due to non-communicable (chronic) diseases was 88% (78.271.000 population) (5), over the world, 65 million people lived with moderate to severe COPD and it is estimated that nearly 3 million people died of COPD in 2015 (5% of all deaths) (6). Besides; COPD -one of the respiratory system diseases- is ranked 4th among the causes of death over the world (7) and it is estimated that in 2020 it will be ranked 3rd (8).

Drug administration, an important nursing role, is a process that includes many disciplines. This process starts with patients' medical examination and physicians' prescription and includes phases of registration, observation of correct reactions and realization of the medical treatment by nurses, physicians, patient himself or his/her significant others (9). Training patients and families about treatment regime, observing patient's response to treatment and success of treatment are too among nurses' responsibilities (10).

According to the studies done in literature; the study of Choi and ChoChung (2001) explored a positive rise in adequacy of MDI among 101 asthma patients after the MDI training session given, the study of Press et al. (2012) was done with 80 COPD patients about adequacy of MDI and 82% of the participants performed steps of MDI use wrongly before the training while 25% of the participants performed the same steps wrongly after the training, the study of Işık et al. (2014) determined mistakes in using inhaler drugs and reported that patients were unable to receive effective and sufficient dose of drugs and the study Özkan and Kaşıkçı (2015) identified mistakes in using MDI and emphasized the usefulness of the training about MDI.

The study was planned to explore the steps where patients made mistakes while using MDI, to find out to what extent they used MDI correctly and to assess the effect of video-training-session upon adequacy of metered dose inhaler (MDI) among individuals with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Those who were voluntary to join the study, were ≥18 years old, had no hearing, vision and speaking impairment, no mental confusion, had full consciousness and orientation, had COPD diagnosis for ≥6 months and used MDI for more than 3 months were included in the study.

Exclusion Criteria:

* Patients who did not volunteer to participate in the study, ≤18 years of age, hearing, vision and speech impairment, mental confusion, without full consciousness and orientation, diagnosed with COPD for less than 6 months and using MDI less than 3 months were not included in the study.

Ages: 48 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
In order to determine the effect of repeated video-training-session method on the adequacy of metered dose inhaler in individuals with COPD, on the 1st day/scores of the 1st and 2nd measurements | one day
  On the 1st day, the 1st measurement was determined by filling out the "MDI Skill Evaluation Form" while the patients were using the MDI sample that did not contain active agent. Next, MDI use was explained through the video twice. After each video and explanation, the patients were asked to use the same MDI sample for 10 minutes. Simultaneously, steps were marked by the researcher through observation on the form, obtaining the scores of the 2nd measurement. The form including 10 adequacy steps about how to use an MDI. According to the scoring system, "0" point refers to a step being performed incorrectly or skipped, while "1" point refers to a correctly performed. The max. score that can be obtained is "10" and the min. score is "0". A total score of 7-10 was assessed as satisfactory, a score of 4-6 as moderate, and a score of 0-3 as unsatisfactory.

SECONDARY OUTCOMES:
In order to determine the effect of repeated video-training-session method on the adequacy of metered dose inhaler in individuals with COPD, on the 2nd day/scores of the 3rd and 4rd measurements | one day
  On the 2nd day, the patients were visited and were again asked to use the metered dose inhaler. While they were using the metered dose inhaler, the "Metered Dose Inhaler Skill Evaluation Form" was marked and "the scores of the 3rd measurement" were found. Later, a video session was held the same way as on the first day, the video was watched twice, and after each repetition the patients were requested to use the metered dose inhaler again. While they were using the metered dose inhaler, the skills and steps were simultaneously marked on the "Metered Dose Inhaler Skill Evaluation Form" and "the scores of the 4th measurement" were determined.

OTHER OUTCOMES:
In order to determine the effect of repeated video-training-session method on the adequacy of metered dose inhaler in individuals with COPD,on the 3rd day/final or 5th measurement | one day
  On the 3rd day, the patients were asked to use an metered dose inhaler that is used in their treatments while the "Metered Dose Inhaler Skill Evaluation Form" was marked and the final measurement was obtained.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Batman Regional State Hospital, Batman
  - Mersin University, Mersin

IPD SHARING:
Plan to Share IPD: No